CLINICAL TRIAL: NCT02864732
Title: A Comparison Between Stabilization Exercises and Stabilization Exercises Supplemented With Neuromuscular Electrical Stimulation: A Feasibility Study
Brief Title: Stabilization Exercises Alone vs Stabilization Exercises Plus Neuromuscular Electrical Stimulation in People With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Saudi Arabian Cultural Mission (Unknown); King Fahad Specialist Hospital Dammam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO12100651
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2017-10

CONDITIONS: Low Back Pain
Keywords: Low back pain; stabilization exercises; neuromuscular electrical stimulation
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Therapy; Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stabilization exercises (Experimental): The stabilization exercises program will consist of exercises for the lower back and abdomen. These exercises include various types of abdominal bracing and bridging and side bridging. The exercises will be performed in supine, sidelying, and quadruped. It involves activation of muscles, dissociation of lumbar spine movement from extremities movement and endurance.
  Interventions: Other: Rehabilitation exercises
- Stabilization exercises plus electrical stimulation (Experimental): The neuromuscular electrical stimulation is a hand-size unit that has four plastic adhesive electrical conductors known as electrodes. These electrodes are going to be placed on the skin covering the lower back muscles. They will deliver an electric current that will generate muscle contraction that resembles normal muscle contraction. This treatment will be given in addition to the stabilization exercise program.
  Interventions: Other: Rehabilitation exercises; Device: Electrical Stimulation

INTERVENTIONS:
Other: Rehabilitation exercises
Device: Electrical Stimulation
  Other Names: Neuromuscular Electrical Stimulation (NMES)
  Arms: Stabilization exercises plus electrical stimulation

SUMMARY:
The purpose of this study is to investigate the feasibility of applying neuromuscular electrical stimulation on the lumbar spine, to report how tolerable the intervention is, and whether the electrical stimulation improve pain, function and muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 years of age and 60.
* Body Mass Index (BMI) of less than 34.
* Low Back Pain duration of 3 months or greater (chronic).
* Minimum pain level on Numeric Pain Rating Scale (NPRS) is 3 or greater.
* Minimum score of Modified Oswestry Disability Questionnaire (MODQ) is 20 or greater.
* Understands English

Exclusion Criteria:

* Positive nerve root tension signs
* Progressive neurological deficit
* Positive Babinski sign.
* Sensory loss that is not in correspondence with dermatomal distribution or peripheral nerves.
* History of spinal surgery
* History of inflammatory joint disease
* Contraindications to physical exercise including history of cardiac disease or being told by a physician not to engage in physical exercise.
* Contraindications to NMES including cardiac pacemaker or skin allergy to adhesives
* History of metastatic cancer in previous 5 years or present treatment for cancer
* Women who indicate that they are pregnant or plan to become pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Z Alrwaily, PhD, Principal Investigator — University of Pittsburgh; Anthony Delitto, PhD, Study Director — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stabilization Exercises: The stabilization exercises program will consist of exercises for the lower back and abdomen. These exercises include various types of abdominal bracing and bridging and side bridging. The exercises will be performed in supine, sidelying, and quadruped. It involves activation of muscles, dissociation of lumbar spine movement from extremities movement and endurance.
  Rehabilitation exercises
- Stabilization Exercises Plus Electrical Stimulation: The neuromuscular electrical stimulation is a hand-size unit that has four plastic adhesive electrical conductors known as electrodes. These electrodes are going to be placed on the skin covering the lower back muscles. They will deliver an electric current that will generate muscle contraction that resembles normal muscle contraction. This treatment will be given in addition to the stabilization exercise program.
  Rehabilitation exercises
  Electrical Stimulation
Period: Overall Study
Arm/Group | Stabilization Exercises | Stabilization Exercises Plus Electrical Stimulation
Started | 15 | 15
Completed | 13 | 13
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: Chronic Low Back Pain Patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Stabilization Exercises | Stabilization Exercises Plus Electrical Stimulation | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.33 (11.3) | 33.40 (9.0) | 35.87 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 4 | 7 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 9 | 13 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.89 (3.9) | 26.47 (2.9) | 26.18 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Electrical Stimulation (NMES)
Description: NMES tolerability was performed by asking each subject in the stab + NMES group to describe their subjective perception of both the intensity and discomfort of the NMES current using the descriptors listed in a table. The descriptors represent two distinct domains of adjectives: the sensory aspect of the perceived intensity of stimulation and the affective aspect of the perceived discomfort. Each aspect has 15 adjectives. Each subject was asked to describe the current using the descriptors listed for each aspect at baseline and at 6 weeks.
  To analyze the the subjects description of the current, the 15 descriptors of each aspect were divided into 3 zones (high, medium, low). The top 5 descriptors in each aspect were considered high, the middle 5 descriptors were considered medium, and the bottom descriptors were considered low.
  Descriptive statistics were used to compare the subjects description of each aspect at baseline and at 6 weeks follow-up.
Time Frame: Participants were followed from baseline to 6 weeks
Population: This outcome measure was only used with the Stabilization plus Electrical Stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Stabilization Exercises Plus Electrical Stimulation
Number analyzed (Participants) | 13
Participants
  Baseline sensory low | 0
  Baseline sensory medium | 5
  Baseline sensory high | 8
  6 week sensory low | 0
  6 week sensory medium | 3
  6 week sensory high | 10
  Baseline discomfort low | 13
  Baseline discomfort medium | 0
  Baseline discomfort high | 0
  6 week discomfort low | 13
  6 week discomfort medium | 0
  6 week discomfort high | 0

2. Primary Outcome: Modified Oswestry Disability Questionnaire (MODQ)
Description: The MODQ is a self-reported measure of disability consisting of 10 domains of functional activities related to low back pain. The domains include pain intensity, personal care, lifting, walking, standing, sitting, traveling, social life, employment/homemaking, and sleeping. Each domain is rated from 0 - 5. The total of all the domains range from 0 - 50. The scores can be multiplied by 2 to get a percentage of functional disability. The higher the percentage the higher the disability.
Time Frame: Baseline to 6 weeks (post-treatment) to 10 weeks (follow up).
Measure: Mean (Standard Deviation); unit: percentage of functional disability
Arm/Group | Stabilization Exercises | Stabilization Exercises Plus Electrical Stimulation
Number analyzed (Participants) | 13 | 13
percentage of functional disability
  Baseline | 30.80 (10.2) | 30.52 (7.8)
  6 weeks | 12.81 (5.2) | 14.49 (10.2)
  10 weeks | 10.00 (5.6) | 13.24 (8.0)

3. Secondary Outcome: Numeric Pain Rating Scale (NPRS)
Description: The NPRS measures pain intensity on an 11-point scale from 0 (no pain) to 10 (maximum pain). The higher the score the worst the pain intensity
Time Frame: Baseline to 6 weeks (post-treatment) to 10 weeks (follow-up)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stabilization Exercises | Stabilization Exercises Plus Electrical Stimulation
Number analyzed (Participants) | 13 | 13
units on a scale
  Baseline | 4.44 (1.8) | 4.20 (1.9)
  6 weeks | 2.07 (1.1) | 2.34 (1.5)
  10 weeks | 1.63 (1.0) | 2.34 (1.5)

4. Secondary Outcome: Fear-avoidance Behavior Questionnaire
Description: The Fear-avoidance Behavior Questionnaire (FABQ) measure avoidant behavior to physical activity or work due to fear of pain. The has two sub scales: physical activity and work. This FABQ consists of 16 items; 5 items for the physical activity sub scale and 11 items for the work subscale. Each item is scored from 0-6. Higher scores on the FABQ are indicative of greater fear and avoidance beliefs. The total score on the FABQ is 66, however, this score is considered separately. The FABQ-physical activity sub scale ranges from 0 - 24 points and the FABQ-work activity ranges from 0 - 42 points.
Time Frame: Baseline to 6 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stabilization Exercises | Stabilization Exercises Plus Electrical Stimulation
Number analyzed (Participants) | 13 | 13
units on a scale
  FABQ-PA Baseline | 12.33 (5.5) | 14.27 (6.5)
  FABQ-PA 6 weeks | 8.41 (6.0) | 10.75 (4.7)
  FABQ-W Baseline | 12.20 (10.9) | 11.67 (10.5)
  FABQ-W 6 weeks | 8.87 (9.6) | 10.75 (7.6)

5. Secondary Outcome: Paraspinal Muscle Strength
Description: The paraspinal muscle strength was assessed using the Biodex 3 Pro dynamometer (20 Ramsey Rd, Shirley, NY 11967). Active extension of the trunk was performed with the subject in a semi-standing position; the subject's hips were flexed at 60 degrees with the feet resting on an adjustable footrest. The thighs were secured to the seat with two Velcro straps. The scapulae rested against a roll that is attached to the chair arms. The trunk was secured with two Velcro straps that crossed the front trunk forming the shape of an X. The subject was asked to extend the trunk by exerting maximal isometric contraction for 5 seconds against the scapular roll. The average of three 5-second trials was recorded. All subjects received the same verbal instruction: "Push your trunk against the scapular roll as strong as you can". The higher the score the stronger the muscles. The range starts from 0 without a limit to the amount of force that could be exerted.
Time Frame: Baseline - 6 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | Stabilization Exercises | Stabilization Exercises Plus Electrical Stimulation
Number analyzed (Participants) | 13 | 13
Nm
  Baseline | 117.29 (57.7) | 154.49 (59.1)
  6 weeks | 162.30 (55.2) | 175.80 (58.4)

6. Secondary Outcome: Patient Satisfaction Survey
Description: Satisfaction level with the interventions. Subjects were asked rate their satisfaction with the treatment by choosing one of the following statements:
  Very satisfied Satisfied Neutral Unsatisfied Very unsatisfied
Time Frame: only post-treatment at 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Stabilization Exercises | Stabilization Exercises Plus Electrical Stimulation
Number analyzed (Participants) | 13 | 13
Participants
  Very satisfied | 10 | 8
  Satisfied | 3 | 5
  Neutral | 0 | 0
  Unsatisfied | 0 | 0
  Very Unsatisfied | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Participants were monitored only for the following select adverse events: a. severe episode of low back pain or b. skin reaction due to use of adhesives.
Arm/Group | Stabilization Exercises | Stabilization Exercises Plus Electrical Stimulation
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
small sample size and no blinding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No